CLINICAL TRIAL: NCT04081051
Title: Impact of Improved Diagnostic Tools, Training and Communication on Acute Fever Case Management and Antibiotic Prescriptions for Children and Adolescents Presenting at Outpatient Facilities in Lower & Middle-Income Countries.
Brief Title: Advancing Access to Diagnostic Innovation Essential for UHC and AMR Prevention
Acronym: Accelerator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University of Oxford (Other); Indian Council of Medical Research (Other Government); WHO, Special Programme for Research and Training in Tropical Diseases (TDR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AM 001
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Acute Febrile Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Diagnostic algorithm( paper and electronic) utilizing pathogen specific and non-pathogen specific point of care, rapid diagnostic tests, behavioral change training for healthcare workers
  Interventions: Other: diagnostic algorithm+Point of care rapid diagnostic tests+ Behavior change ( assessed together as a single package of interventions)
- control (No Intervention): Standard of care practices for acute febrile illness

INTERVENTIONS:
Other: diagnostic algorithm+Point of care rapid diagnostic tests+ Behavior change ( assessed together as a single package of interventions) — Diagnostic algorithm utilizing pathogen specific and non-pathogen specific point of care, rapid diagnostic tests, behavioral change intervention for healthcare workers
  Arms: Intervention

SUMMARY:
This study aims to evaluate clinical outcomes and antibiotic prescription patterns following the use of diagnostic algorithms, point of care (PoC) rapid diagnostic tests, and behaviour change interventions in cases of acute febrile illnesses in children, adolescents and adults presenting at out patient clinics in lower and middle income countries. The study is to be implemented in 2 phases- the first run from 2020 to 2021 and the 2nd phase from 2021 to 2022 to include COVID-19 PoCTs.

DETAILED DESCRIPTION:
Background and rationale. 'Just-in-case' antibiotic prescribing practices is one of the causes of inadequate management of 'acute febrile illnesses' and AMR in Low- and Middle-income Countries (LMICs). At the same time, some people who would require antibiotic treatment do not get it. An improvement in case management and prescription practice might lead to a decrease in morbidity and mortality. Success will mean making significant steps toward achieving the dual goal of improving UHC and tackling AMR.

The PICO question addressed is: in children/ adolescents and adults (Population) presenting to outpatient clinics / peripheral health centres in LMICs with acute febrile illness/Respiratory Tract Infection can a combination of available PoC rapid diagnostic tests, diagnostic aids/algorithms, clinic process flow and, training and communication (Intervention) improve management of acute febrile illnesses and better target the use of antibiotics / reduce unnecessary antibiotic prescriptions (Outcomes) compared to current practice (Control)?

Primary objective(s).

To evaluate the impact of a package of interventions (point of care [PoC] tests, clinical algorithm, clinic process flow, training and communication tools) on clinical outcomes and antibiotic prescriptions, with standard-of-care practices, in children and adolescents presenting with acute febrile illnesses (defined as fever with no focus or Respiratory Tract Infection lasting for no more than 7 days), at outpatient clinics.

Secondary objective(s)

1. To improve the management of acute febrile illness
2. To promote rational and targeted use of antibiotics for acute febrile illness
3. To determine the aetiology of fever in patients presenting to outpatient facilities using available PoC diagnostic tests
4. To study the safety and feasibility of a package of interventions compared to current practice of care
5. To assess the effectiveness of training and communication tools to adherence to the prescribed treatment

Primary endpoints

1. Proportion of outpatient cases of acute febrile illness with favourable outcome (defined as being alive and asymptomatic).
2. antibiotic prescriptions rates for acute febrile illness in the clinic Secondary endpoints (outcomes) 1. Duration of time spent in the clinic

2. Proportion of patients treated for specific bacterial infection 3. Proportion of patients with disease specific diagnosis identified by PoC tests 4. Frequency of serious adverse event (SAE) within 7 days of recruitment 5. Frequency of unscheduled (unplanned) visit within 7 days of recruitment 6. Training and communication package uptake 7. Proportion of patients prescribed antibiotic at clinic who reported adherence to prescription on day 7 8. Proportion of patients who were not prescribed antibiotics at clinic who received antibiotics elsewhere between day 0 and day 7 9. Behaviour Change Intervention Recommendations

Trial design: A multi-centre, open label, two arm, randomized-controlled trial

Trial sites: This study will be conducted in outpatient departments and primary care clinics in Burkina Faso, Ghana, India, Nepal and Uganda.

Trial population: The study population will consist of children, adolescents and adults presenting to the health care facility, or provider, with acute fever or history of fever

Sample Size: 19,922

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with fever with no focus/RTI:

  * Children (6 months to <12 years) and adolescents (12 years to less than 18 years old) of both sexes .
  * Presenting with an acute febrile illness defined as temperature of >37.5°C or history of fever within the last 7 days with no focus or suspected RTI.
  * Parent/guardian providing written informed consent for their children if less than 18 years of age.
  * Obtain assent for adolescent between 12 and less than 18 years old
  * Willing to provide blood and other samples and adhere to study procedures explained in the consent forms following the protocol.
  * Available and willing to return for follow-up visit at the health facility on day 7 (+/- 2 days).

Exclusion Criteria:

* o Children and adolescents from 6 months to less than 18 years old presenting with chronic febrile illness (fever lasting more than 7 days).

  * Patients with acute febrile illness outside the allowed age range for the site.
  * Severely ill patients requiring hospital admission or referral as assessed by the study clinicians.
  * Anyone refusing consent to the study or not able to attend the health centre for follow-up (adults, the children of parents/guardians, or adolescents who refuse or are missed when asking for consent).

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17294 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of acute febrile cases with favorable clinical outcomes at day 7 | Day 7
  Favorable defined as being alive and asymptomatic.
Antibiotic prescription rates in acute fever cases | Day 0
  Proportion of antibiotic prescriptions for acute febrile illness in the clinic

SECONDARY OUTCOMES:
Proportion of participants with acute fever Diagnoses identified by point of care tests. | Day 0
  Proportion of patients with disease specific diagnosis identified by PoC tests
Adverse events | Day 7
  Frequency of adverse events within 7 days of recruitment
Time spent in the clinic | Day 0
  Time spent in the clinic
Proportion of study participants who adhered to antibiotic prescriptions | Day 7
  Adherence to antibiotic prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Piero Olliaro, MD, Study Director — Foundation for Innovative New Diagnostics (FIND)
Locations (8):
- IRSS-DRCO/Clinical Research Unit of Nanoro (CRUN), Nanoro, Burkina Faso
- Shai-Osudoku District Hospital, Accra, Dodowa, Ghana
- India (4):
  - Jan Swathya Sahyog, Ganiyari, Chhattisgarh
  - National Institute of Cholera & Enteric Diseases, Beliaghata, Kolkata
  - R D Gardi Medical College, Ujjain, Madhya Pradesh
  - Post Graduate Insitute Medical Education and Research, Chandigarh
- Patan Academy of Health Sciences, Lalitpur, Lagankhel, Nepal
- Infectious Disease research collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
to be discussed

REFERENCES:
- [Derived] Kiemde F, Nkeramahame J, Ibarz AB, Dittrich S, Olliaro P, Valia D, Rouamba T, Kabore B, Kone AN, Sawadogo S, Bere AW, Some DY, Some AM, Compaore A, Horgan P, Weber S, Keller T, Tinto H. Impact of a package of point-of-care diagnostic tests, a clinical diagnostic algorithm and adherence training on antibiotic prescriptions for the management of non-severe acute febrile illness in primary health facilities during the COVID-19 pandemic in Burkina Faso. BMC Infect Dis. 2024 Aug 27;24(1):870. doi: 10.1186/s12879-024-09787-y. PMID 39192209
- [Derived] Adjei A, Kukula V, Narh CT, Odopey S, Arthur E, Odonkor G, Mensah MM, Olliaro P, Horgan P, Dittrich S, Moore CE, Salami O, Awini E, Nkeramahame J, Williams J, Baiden R. Impact of Point-of-Care Rapid Diagnostic Tests on Antibiotic Prescription Among Patients Aged <18 Years in Primary Healthcare Settings in 2 Peri-Urban Districts in Ghana: Randomized Controlled Trial Results. Clin Infect Dis. 2023 Jul 25;77(Suppl 2):S145-S155. doi: 10.1093/cid/ciad328. PMID 37490745
- [Derived] Kiemde F, Valia D, Kabore B, Rouamba T, Kone AN, Sawadogo S, Compaore A, Salami O, Horgan P, Moore CE, Dittrich S, Nkeramahame J, Olliaro P, Tinto H. A Randomized Trial to Assess the Impact of a Package of Diagnostic Tools and Diagnostic Algorithm on Antibiotic Prescriptions for the Management of Febrile Illnesses Among Children and Adolescents in Primary Health Facilities in Burkina Faso. Clin Infect Dis. 2023 Jul 25;77(Suppl 2):S134-S144. doi: 10.1093/cid/ciad331. PMID 37490742
- [Derived] Compaore A, Ekusai-Sebatta D, Kaawa-Mafigiri D, Kukula V, Odopey S, Kapisi J, Hopkins H, Kiemde F, Tinto H, Baiden R, Olliaro P, Nkeramahame J, Dittrich S, Horgan P; ADIP study group. Viewpoint: Antimicrobial Resistance Diagnostics Use Accelerator: Qualitative Research on Adherence to Prescriptions. Clin Infect Dis. 2023 Jul 25;77(Suppl 2):S206-S210. doi: 10.1093/cid/ciad323. PMID 37490738
- [Derived] Salami O, Horgan P, Moore CE, Giri A, Sserwanga A, Pathak A, Basnyat B, Kiemde F, Smithuis F, Kitutu F, Phutke G, Tinto H, Hopkins H, Kapisi J, Swe MMM, Taneja N, Baiden R, Dutta S, Compaore A, Kaawa-Mafigiri D, Hussein R, Shakya SU, Kukula V, Ongarello S, Tomar A, Chadha SS, Walia K, Kelly-Cirino C, Olliaro P. Impact of a package of diagnostic tools, clinical algorithm, and training and communication on outpatient acute fever case management in low- and middle-income countries: protocol for a randomized controlled trial. Trials. 2020 Nov 25;21(1):974. doi: 10.1186/s13063-020-04897-9. PMID 33239106